CLINICAL TRIAL: NCT00795938
Title: An Open-Label, Crossover Study In Healthy Volunteers To Evaluate The Pharmacokinetics Of Sildenafil Following Administration Of An Experimental Tablet Of Sildenafil With Or Without Water Relative To Viagra® Conventional Oral Tablet With Water.
Brief Title: Study to Compare the Blood Levels of Sildenafil Following Administration of an Experimental Tablet vs. the Conventional Oral Tablet in Healthy Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A1481266
Record Dates: First submitted 2008-11-19; First posted 2008-11-21 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Conventional Oral Tablet With Water (Active Comparator)
  Interventions: Drug: Sildenafil
- Experimental Tablet With Water (Experimental)
  Interventions: Drug: Sildenafil
- Experimental Tablet Without Water (Experimental)
  Interventions: Drug: Sildenafil

INTERVENTIONS:
Drug: Sildenafil — Single Dose of 50 mg Sildenafil Oral Tablet With Water
  Arms: Conventional Oral Tablet With Water
Drug: Sildenafil — Single Dose of 50 mg Sildenafil Experimental Tablet With Water
  Arms: Experimental Tablet With Water
Drug: Sildenafil — Single Dose of 50 mg Sildenafil Experimental Tablet Without Water
  Arms: Experimental Tablet Without Water

SUMMARY:
This study to will compare the blood levels of sildenafil following administration of an experimental tablet vs. the conventional oral tablet.

ELIGIBILITY:
Inclusion Criteria:

Healthy males between the ages of 18 and 55 years. Body Mass Index of 18 to 30 kg/m2, and a total body weight >50 kg (110 lbs).

Exclusion Criteria:

Smoking in excess of the equivalent of 5 cigarettes per day. Treatment with an experimental drug within 30 days or sildenafil, vardenafil, tadalfil within 4 days before first study dose.

Develop blood pressure lowering or experience dizziness, lightheadedness when going from the laying down position to standing position.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2008-10; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Blood levels of sildenafil | 1 day

SECONDARY OUTCOMES:
Blood levels of a metabolite of sildenafil | 1 day
Safety | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States